CLINICAL TRIAL: NCT04553237
Title: Clinical Prognosis After Stroke in Nonagenarian Patients Treated With Thrombolysis or Mechanical Thrombectomy
Acronym: PCAT
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PCAT
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients over 90 years old
- Patients between 70 and 89 years of age.

SUMMARY:
Stroke is a significant cause of death and disability in France and internationally. The incidence of stroke increases with age, equal for both sexes. Of all strokes, 50% of cases occur in patients over 75 years of age. This advanced age leads to a high risk of mortality, long hospitalization, causing neurological sequelae in most cases.

Neurological handicap in the elderly is due to a high rate of comorbidity, reduced neuronal plasticity, nutritional status, and the short time to convert the penumbra area to ischemia.

Currently the standard treatment for the acute phase of HF is thrombolysis or thrombectomy.

The principle of thrombolysis is based on the use of a thrombolytic drug (Actylise®). It is a tissue plasminogen activator (t-PA) that will cause lysis and dissolution of clots blocking the artery. Thrombolysis is recommended until 4:30 a.m. after the onset of symptoms in the absence of contraindication.

Mechanical thrombectomy consists of removing the blood clot by introducing a probe into the artery having a proximal carotid or sylvic occlusion in its M1 portion or in the vertebro-basilar territory of an indeterminate schedule of less than 24 hours or determined from 6 hours to 24 hours having a radio-clinical mismatch, according to the DAWN study. The results of this study were analyzed according to age, NIHSS score and lesion volume on perfusion scanner or MRI (RAPID software). The interim analysis at 31 months on 206 randomized patients (107 thrombectomies versus 99 medical treatments alone) showed a clear superiority of the thrombectomy, leading to the premature end of the study, over the handicap at 3 months with more than 35 % of independent patients.

In most of the randomized studies, patients over 90 years of age have been excluded or are under-represented. This lack of data therefore does not make it possible to determine the effectiveness of thrombolysis or thrombectomy treatments in these patients.

A recent meta-analysis has shown that the functional recovery in these patients treated by thrombectomy is superior to those of the same age without thrombectomies. According to American studies, the advanced age of a patient is not a contraindication to this treatment.

Patients affected by a cerebral infarction represent 40 to 50% of hospitalizations in the neurology department of the Groupe Hospitalier Paris Saint-Joseph. In the intensive care of the neuro-vascular unit, the patient is received as quickly as possible to decide whether he can benefit from an extreme emergency treatment (intravenous thrombolysis or thrombectomy).

The present study should show that the clinical course after treatment in patients over 90 years of age is substantially comparable to younger patients, and that age is not a contraindication to treatment in the acute phase of stroke in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 70 years old
* Patient treated in the neurology department of Paris Saint-Joseph hospital for a stroke between 2017 and 2019
* Patient treated by thrombolysis less than 4:30 after the onset of symptoms and / or by mechanical thrombectomy less than 24 hours.
* French-speaking patient

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under legal protection
* Patient objecting to the use of their data for this research

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients treated for stroke in the neurology department within the Groupe Hospitalier Paris Saint Joseph, between January 01, 2017 and December 31, 2019, i.e. 122 patients.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Management of stroke between two groups of patients. | Day 90
  This outcome corresponds to the comparaison of functional recovery at D90 after a stroke as measured by the Modified Rankin scale for measuring the degree of disability or dependence in the daily activities of patients.
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.

SECONDARY OUTCOMES:
Symptomatic hemorrhagic changes | Day 90
  This outcome corresponds to the rate of patients with hemorrhagic transformation.
Intra-hospital mortality | Day 90
  This outcome corresponds to the rate of patients with in-hospital mortality.
Other complications | Day 90
  This outcome corresponds to the rate of patients presenting others complications during hospitalisation.

CONTACTS AND LOCATIONS:
Overall Officials: IOANA BABICIU, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Result] Murphy SL, Xu J, Kochanek KD, Curtin SC, Arias E. Deaths: Final Data for 2015. Natl Vital Stat Rep. 2017 Nov;66(6):1-75. PMID 29235985
- [Result] Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, Biller J, Brown M, Demaerschalk BM, Hoh B, Jauch EC, Kidwell CS, Leslie-Mazwi TM, Ovbiagele B, Scott PA, Sheth KN, Southerland AM, Summers DV, Tirschwell DL; American Heart Association Stroke Council. 2018 Guidelines for the Early Management of Patients With Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2018 Mar;49(3):e46-e110. doi: 10.1161/STR.0000000000000158. Epub 2018 Jan 24. PMID 29367334
- [Result] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Result] Saposnik G, Cote R, Phillips S, Gubitz G, Bayer N, Minuk J, Black S; Stroke Outcome Research Canada (SORCan) Working Group. Stroke outcome in those over 80: a multicenter cohort study across Canada. Stroke. 2008 Aug;39(8):2310-7. doi: 10.1161/STROKEAHA.107.511402. Epub 2008 Jun 12. PMID 18556583
- [Result] Castonguay AC, Zaidat OO, Novakovic R, Nguyen TN, Taqi MA, Gupta R, Sun CH, Martin C, Holloway WE, Mueller-Kronast N, E English J, Linfante I, Dabus G, Malisch TW, Marden FA, Bozorgchami H, Xavier A, Rai AT, Froehler MT, Badruddin A, Abraham MG, Janardhan V, Shaltoni H, Yoo AJ, Abou-Chebl A, Chen PR, Britz GW, Kaushal R, Nanda A, A Issa M, Nogueira RG. Influence of age on clinical and revascularization outcomes in the North American Solitaire Stent-Retriever Acute Stroke Registry. Stroke. 2014 Dec;45(12):3631-6. doi: 10.1161/STROKEAHA.114.006487. Epub 2014 Oct 30. PMID 25358699
- [Result] Chandra RV, Leslie-Mazwi TM, Oh DC, Chaudhry ZA, Mehta BP, Rost NS, Rabinov JD, Hirsch JA, Gonzalez RG, Schwamm LH, Yoo AJ. Elderly patients are at higher risk for poor outcomes after intra-arterial therapy. Stroke. 2012 Sep;43(9):2356-61. doi: 10.1161/STROKEAHA.112.650713. Epub 2012 Jun 28. PMID 22744644
- [Result] Sharma JC, Fletcher S, Vassallo M. Strokes in the elderly - higher acute and 3-month mortality - an explanation. Cerebrovasc Dis. 1999 Jan-Feb;9(1):2-9. doi: 10.1159/000015889. PMID 9873157
- [Result] Sharobeam A, Cordato DJ, Manning N, Cheung A, Wenderoth J, Cappelen-Smith C. Functional Outcomes at 90 Days in Octogenarians Undergoing Thrombectomy for Acute Ischemic Stroke: A Prospective Cohort Study and Meta-Analysis. Front Neurol. 2019 Mar 20;10:254. doi: 10.3389/fneur.2019.00254. eCollection 2019. PMID 30949120
- [Result] To CY, Rajamand S, Mehra R, Falatko S, Badr Y, Richards B, Qahwash O, Fessler RD. Outcome of mechanical thrombectomy in the very elderly for the treatment of acute ischemic stroke: the real world experience. Acta Radiol Open. 2015 Sep 10;4(9):2058460115599423. doi: 10.1177/2058460115599423. eCollection 2015 Sep. PMID 26445678